CLINICAL TRIAL: NCT04968392
Title: Analgesic Efﬁcacy of Single-shot Adductor Canal Block With Levobupivacaine and Dexmedetomidine in Total Knee Arthroplasty: a Randomized Clinical Trial
Brief Title: Single-shot Adductor Canal Block With Levobupivacaine and Dexmedetomidine in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17300626
Record Dates: First submitted 2021-07-04; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Adductor Canal Block; Levobupivacaine; Dexmedetomidine
Keywords: Dexmedetomidine; levobupivacaine; Adductor Canal Block
MeSH Terms: interventions — Dexmedetomidine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L group (Experimental): 20 mL of 0.25% levobupivacaine plus 1 mL normal saline
  Interventions: Drug: Levobupivacaine
- LD group (Experimental): 20 mL of 0.25% levobupivacaine plus 0.5 µg/kg dexmedetomidine
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — 20 mL of 0.25% levobupivacaine plus 0.5 µg/kg dexmedetomidine
  Arms: LD group
Drug: Levobupivacaine — 20 mL of 0.25% levobupivacaine plus 1 mL normal saline
  Arms: L group

SUMMARY:
Total knee arthroplasty surgery is associated with severe postoperative pain and adequate pain management is necessary for early postoperative mobilization and rehabilitation. Although good postoperative pain control may be achieved by continuous epidural anesthesia or femoral nerve block, both methods have adverse effects such as muscle weakness, which may delay postoperative mobilization.

DETAILED DESCRIPTION:
The adductor canal block (ACB) is a relatively new block providing analgesia for knee surgery, which not only blocks the largest sensory branch of the femoral nerve but also results in less reduction of quadriceps muscle strength, compared with the femoral nerve block (FNB) in adult patients.

Randomized controlled trials have revealed that ACB provides at least equal analgesia as FNB, preserves quadriceps muscle strength better than FNB, and thus allowing for functional recovery within the first 24-hour post-TKA. However, one important limitation of single-shot peripheral nerve block is the short duration of analgesia. Because the average duration of severe pain after TKA takes 2-3 days, a continuous ACB via catheter would seem to be a good choice. Unfortunately, perineural catheters may be technically difficult to insert, are prone to premature dislodgement, and may increase infection risk. There also were some case reports of local anesthetic-induced myotoxicity after continuous ACB.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* undergoing elective primary total knee arthroplasty surgery under spinal anesthesia.

Exclusion Criteria:

* Patients with a known history of significant hepatic,
* renal, heart disease, autoimmune disease,
* any known convulsive disorder, any psychiatric disorders, chronic pain,
* pregnant females, regular use analgesics, anti-depressants, or opioids in the previous 2 months, revision surgery, morbid obesity, allergy to local anesthetics or morphine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
the first analgesia rescue call. | 24 hours postoperative
  time to the first analgesic request.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer MC, Pogatzki-Zahn EM, Zahn PK. Regional analgesia techniques for total knee replacement. Curr Opin Anaesthesiol. 2014 Oct;27(5):501-6. doi: 10.1097/ACO.0000000000000115. PMID 25111605
- [Background] Jaeger P, Koscielniak-Nielsen ZJ, Schroder HM, Mathiesen O, Henningsen MH, Lund J, Jenstrup MT, Dahl JB. Adductor canal block for postoperative pain treatment after revision knee arthroplasty: a blinded, randomized, placebo-controlled study. PLoS One. 2014 Nov 11;9(11):e111951. doi: 10.1371/journal.pone.0111951. eCollection 2014. PMID 25386752
- [Background] Jiang X, Wang QQ, Wu CA, Tian W. Analgesic Efficacy of Adductor Canal Block in Total Knee Arthroplasty: A Meta-analysis and Systematic Review. Orthop Surg. 2016 Aug;8(3):294-300. doi: 10.1111/os.12268. PMID 27627711